CLINICAL TRIAL: NCT04425434
Title: Therapeutic Recommendations For The Treatment Of Children With A Retinoblastoma
Acronym: GFARB12019
Status: Recruiting | Type: Observational
Sponsor: French Africa Pediatric Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: GFAOP RB1
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: OBSERVATIONAL — We will look at the outcome of the the children treated to see if the survival is improved when these therapeutic measures are followed.

SUMMARY:
As the survival of children with retinoblastoma in high income countries is higher than 95% including the bilateral forms this study hopes to improve the outcome in low income countries in Africa by improving early diagnosis and early implementation of this protocol of therapeutic recommendations for treatment.

DETAILED DESCRIPTION:
In this study we will try to improve the outcome for children with stage II disease. It is hoped that we will be able to show that with early intervention correct early diagnosis the survival of these children is greatly improved. The collection of data in this observational study will allow us to show this improvement, by analysis of stage, treatment and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral intraocular Retinoblastoma (RB)
* Unilateral extraocular intraorbital (RB)
* Bilateral intraocular (RB)
* bilateral intraocular (RB) on one side and extraocular but intraorbital on the other side.

Exclusion Criteria:

* Externalized tumor mass
* massive extension to optic nerve up to optical channeltumor
* intracranial extension leptomeninges
* cerebral parenchyma
* extension to regional lymph nodes and/or remote metastases.
* cerebrospinal fluid involvement.
* Trilateral RB
* Incapacity to followed the whole treatement.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: all children presenting at participating units who can be treated
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Number of cases with retinoblastoma in each participating hospital. | 10 years
  Evaluation of the number of cases registered .
Number of cases with stage 2 disease | 10 years
  Evaluation of the number of cases registered with stage 2 disease.
Feasibility of these therapeutic recommendations in an African setting | 10 years
  Evaluate the application of these therapeutic recommendations
Evaluating the treatment given. | 10 years
  Comparison of treatment given and recommended treatment.
follow up | 10 years
  analysis of the number of children alive or dead after treatment

CONTACTS AND LOCATIONS:
Overall Officials: FOUSSEYNI Mr TRAORE, Dr;, Principal Investigator — AMCC AND GFAOP
Locations (7):
- Hopital Yalgado Ouedraogo, Ouagadougou, Burkina Faso
- CHU de Treichville à ABIDJAN, Abidjan, Côte d’Ivoire
- Democratic Republic of the Congo (2):
  - CUK (Cliniques Universitaires de Kinshasa), Kinshasa, Kinshasa City
  - Cliniques Universitaires de Lubumbashi (CUL), Lubumbashi
- HJRA, Hôpital universitaire Joseph Ravoahangy Andrianavalona, Antananarivo, Ampefiloha, Madagascar
- CHU Gabriel Touré (HGT), Bamako, Mali
- Hôpital Aristide Le Dantec,, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No